CLINICAL TRIAL: NCT01841619
Title: Proof-of-Concept Study of IVIg Efficacy in Patients With Cutaneous Lupus Erythematosus
Brief Title: IVIg Efficacy Study to Treat Cutaneous Lupus Erythematosus
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Grifols Therapeutics LLC (Industry)
Responsible Party: Principal Investigator, Sergei Grando, Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-9351
Record Dates: First submitted 2013-04-21; First posted 2013-04-26 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-03

CONDITIONS: Cutaneous Lupus Erythematosus
Keywords: skin, lupus, intravenous immunoglobulin, ivig
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IVIg as a monotherapy (Active Comparator): IVIg will be used as a first line treatment. Topical treatment will be stopped at the beginning of IVIg therapy.
  Interventions: Drug: IVIg

INTERVENTIONS:
Drug: IVIg — All enrolled subjects will receive IVIg treatment following the protocol that proved to be efficacious in the treatment of patients with autoimmune blistering diseases as well as some patients with CLE. The drug will be administered at 500 mg/kg/day on consecutive days up to a total of 2 g/kg/month for 3 months in the Institute for Clinical and Translational Science (ICTS) at University of California, Irvine. After 3 months of treatment, IVIg will be discontinued and the subjects will be monitored for additional 6 months for a possible relapse. In the case of relapse, which is expected to occur in <25% subjects, the subjects will be re-treated by the standard protocol.
  Other Names: Intravenous Immunoglobin

SUMMARY:
The purpose of this research study is to show that non-steroidal treatment with intravenous immunoglobulin (IVIg) can replace current systemic immunosuppressive therapy in cutaneous lupus erythematosis (CLE) patients.

DETAILED DESCRIPTION:
The ultimate goal of this pilot project is to generate proof-of-concept data showing that treatment with intravenous immunoglobulin (IVIg) can replace current systemic immunosuppressive therapy in cutaneous lupus erythematosis (CLE) patients. This project has relevant clinical implications due to the severe side effects of and lack of response to current therapies.

From the review of literature, it can be postulated that:

1. the beneficial effects of IVIg for patients with CLE should be prompt, with marked improvement within a few weeks;
2. clinical improvement should last several weeks after the last infusion; and
3. remission may be prolonged by maintenance IVIg therapy.

Although this is only a non-controlled study, the investigator expects that IVIg will improve CLE, including those resistant to standard treatments. It is anticipated that treatment with IVIg will facilitate healing of extensive cutaneous lesions and achieve rapid remission. Maintenance therapy with repeated monthly pulses of IVIg is expected to keep the disease in remission during the treatment-free follow up observational period. The results will provide the basis a multicenter randomized controlled study to identify which CLE subsets will benefit the most and which protocol will provide the optimal clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Be at least 18 years of age at time of informed consent.
* Have had a diagnosis of CLE
* Currently has active CLE (any subtype) established by standard clinical and histo- and immunopathologic criteria
* Falls into one of the two following cohorts:
* Cohort 1 - Has received a standard systemic therapy without a therapeutic response for a minimum of one month
* Cohort 2 - Has not received any systemic treatment

Exclusion Criteria:

* Subject is not over 18 years of age.
* Subject cannot understand or follow directions.
* Subject is a female of child-bearing potential and unwilling to use a form of highly effective birth control.
* Subject is pregnant, planning to get pregnant, or breast feeding.
* Subject has a known history of immunoglobulin A (IgA) deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergei Grando, MD PhD D.Sc., Principal Investigator — University of California, Irvine
Locations (2):
- United States (2):
  - The Institute for Clinical and Translational Science (ICTS), Irvine, California
  - Unversity of California, Irvine Healthcare, Dermatology, Gottschalk Medical Plaza, Irvine, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IVIg as a Monotherapy
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IVIg as a Monotherapy
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 1

OUTCOME MEASURES:

1. Secondary Outcome: Mean Percent Change in Physician's Subjective Assessment of Improvement (PSAI)
Description: At clinic visits, the investigator will categorize the change in disease activity in each patient as improved, unchanged, or worse since the last visit. Estimated change in disease activity will be based on the investigator's subjective assessment of the patient's skin disease.
  Results expressed relative to the mean initial value of all patients, taken as 100%. Each proceeding visit will be relative to the initial visit. A decrease in percentage represents improvement while an increase in percentage indicates worsening of CLE. Visits occur on a month-to-month basis.
Time Frame: Initial, 1st Visit - 9th Visit
Measure: Mean (Standard Deviation); unit: Percent of Baseline
Arm/Group | IVIg as a Monotherapy
Number analyzed (Participants) | 16
Percent of Baseline
  Intial | 100 (0)
  1st Visit | 100 (0)
  2nd Visit | 100 (0)
  3rd Visit | 136 (79)
  4th Visit | 104 (48)
  5th Visit | 105 (52)
  6th Visit | 117 (37)
  7th Visit | 133 (47)
  8th Visit | 150 (77)
  9th Visit | 100 (29)

2. Secondary Outcome: Mean Percent Change in Physician's Subjective Assessment of Severity (PSAS)
Description: as for outcome 1
Time Frame: Initial, 1st Visit - 9th Visit
Measure: Mean (Standard Deviation); unit: Percent of Baseline
Arm/Group | IVIg as a Monotherapy
Number analyzed (Participants) | 16
Percent of Baseline
  Initial | 100 (0)
  1st Visit | 100 (0)
  2nd Visit | 98 (8)
  3rd Visit | 100 (10)
  4th Visit | 97 (18)
  5th Visit | 92 (19)
  6th Visit | 92 (18)
  7th Visit | 92 (20)
  8th Visit | 90 (18)
  9th Visit | 90 (17)

3. Primary Outcome: Cutaneous Lupus Erythematosus Disease Area and Severity Index - Total Activity Score (CLASI - TAS)
Description: Disease activity will be measured using the CLASI activity score that describes the activity of the disease. This score ranges from 0-70, with higher scores indicating more severe skin disease. This clinical assessment tool enables standardized assessments of response to therapy.
  Results expressed relative to the mean initial value of all patients, taken as 100%. Each proceeding visit will be relative to the initial visit. A decrease in percentage represents improvement while an increase in percentage indicates worsening of CLE. Visits occur on a month-to-month basis.
Time Frame: Initial, 1st Visit - 9th Visit
Measure: Mean (Standard Deviation); unit: Percent of Baseline
Arm/Group | IVIg as a Monotherapy
Number analyzed (Participants) | 16
Percent of Baseline
  Initial | 100 (0)
  1st Visit | 94 (30)
  2nd Visit | 84 (29)
  3rd Visit | 94 (52)
  4th Visit | 86 (19)
  5th Visit | 85 (14)
  6th Visit | 72 (37)
  7th Visit | 68 (33)
  8th Visit | 81 (17)
  9th Visit | 71 (13)

4. Secondary Outcome: Cutaneous Lupus Erythematosus Disease Area and Severity Index - Total Damage Score (CLASI - TDS)
Description: Disease activity will be measured using the CLASI activity score that describes the damage of the disease. This score ranges from 0-70, with higher scores indicating more severe skin disease. This clinical assessment tool enables standardized assessments of response to therapy.
  Results expressed relative to the mean initial value of all patients, taken as 100%. Each proceeding visit will be relative to the initial visit. A decrease in percentage represents improvement while an increase in percentage indicates worsening of CLE. Visits occur on a month-to-month basis.
  All patients were measured identically in all visits.
Time Frame: Initial, 1st Visit - 9th Visit
Measure: Mean (Standard Deviation); unit: Percent of Baseline
Arm/Group | IVIg as a Monotherapy
Number analyzed (Participants) | 16
Percent of Baseline
  Initial | 100 (0)
  1st Visit | 100 (0)
  2nd Visit | 100 (0)
  3rd Visit | 100 (0)
  4th Visit | 100 (0)
  5th Visit | 100 (0)
  6th Visit | 100 (0)
  7th Visit | 100 (0)
  8th Visit | 100 (0)
  9th Visit | 100 (0)

5. Primary Outcome: Skindex 29
Description: The subjects also evaluated their skin-specific quality of life with the Skindex-29 - the questionnaire consisting of 29 items used to calculate three subscales: symptoms (pain, itch, burning, sensitivity), emotions (depression, anxiety, embarrassment, anger) and functioning (sleep, relationships with others). All assessments were repeated at all study visits. Results expressed relative to the mean initial value of all patients, taken as 100%. Each proceeding visit will be relative to the initial visit. A decrease in percentage represents improvement while an increase in percentage indicates worsening of CLE. Visits occur on a month-to-month basis.
Time Frame: Initial, 1st Visit - 9th Visit
Measure: Mean (Standard Deviation); unit: Percent of Baseline
Arm/Group | IVIg as a Monotherapy
Number analyzed (Participants) | 16
Percent of Baseline
  Initial | 100 (0)
  1st Visit | 97 (3)
  2nd Visit | 94 (9)
  3rd Visit | 92 (12)
  4th Visit | 90 (15)
  5th Visit | 81 (21)
  6th Visit | 79 (23)
  7th Visit | 83 (30)
  8th Visit | 99 (11)
  9th Visit | 82 (21)

ADVERSE EVENTS:
Arm/Group | IVIg as a Monotherapy
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 9/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVIg as a Monotherapy (N=16)
Anemia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Headache (Nervous system disorders) | 3 (5)
Oral Lupus Flare (Immune system disorders) | 1
Back Spasms (Musculoskeletal and connective tissue disorders) | 1
Diabetic Foot Ulcer (Infections and infestations) | 1
Herpes - Associated Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1
Lupus Flare (Immune system disorders) | 2
GI Upset (Gastrointestinal disorders) | 1
Fever (General disorders) | 2
Nausea/Vomting (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No